CLINICAL TRIAL: NCT03618979
Title: A Randomized Controlled Trial to Assess the Effects of Autologous Platelet Rich Plasma, Platelet Lysate, and Platelet Poor Plasma on Atrophied Multifidus Muscles in Patients With Axial Lower Back Pain
Brief Title: A Trial Comparing Three Orthobiologic Therapies on Atrophied Multifidus Muscles in Patients With Low Back Pain
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Regenexx, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RGX2018-RCT01
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Low Back Pain
Keywords: regenerative medicine; low back pain; multifidus; platelet rich plasma
MeSH Terms: conditions — Low Back Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PPP treatment (Experimental): Platelet Poor Plasma (PPP) into the multifidus on each side and at each level 1 time per week for 6 weeks (series of 6 injections)
  Interventions: Biological: PPP treatment
- PRP treatment (Experimental): 5x concentration Platelet Rich Plasma (PRP) injected into the multifidus on each side and at each level 1 time per week for 6 weeks (series of 6 injections)
  Interventions: Biological: PRP treatment
- PRP and PL Combo treatment (Experimental): 5x concentration PRP injected into the multifidus, along with a facet joint injection with 14x PRP into each joint and capsule, and transforaminal epidural injection with of 3x concentrated platelet lysate (PL) and 0.5% ropivacaine on each side and at each level 1 time every 2 weeks for 6 weeks total (series of 3 injections)
  Interventions: Biological: PRP and PL Combo treatment

INTERVENTIONS:
Biological: PPP treatment — The day prior to or the morning of the procedure, patient will have their blood drawn by a phlebotomist and processed into 5 or 10 cc of PPP depending on if there is lumbar multifidus atrophy in one or two levels. Using sterile technique and ultrasound guidance, once touching the lamina the physician will inject 2.5 cc of PPP. The physician will then repeat the procedure on the opposite side.
  Arms: PPP treatment
Biological: PRP treatment — The day prior to or the morning of the procedure, patient will have their blood drawn by a phlebotomist and processed into 5 or 10 cc of 5x PRP depending on if there is lumbar multifidus atrophy in one or two levels. Using sterile technique and ultrasound guidance, once touching the lamina the physician will inject 2.5 cc of PRP and remove the needle. The physician will then repeat the procedure on the opposite side and at the next level if indicated.
  Arms: PRP treatment
Biological: PRP and PL Combo treatment — The day prior to or the morning of the procedure patient will have their blood drawn by a phlebotomist and processed into 5 or 10 cc of 5x PRP and 5 or 10 cc of PL and 2 or 4 cc of 14x PRP depending on if there will be one or two levels injected. Using sterile technique, under ultrasound visualization into the lumbar multifidus and onto the lamina, the physician will inject the PRP and remove the needle. Under intermittent x-ray, epidural flow is confirmed with contrast, the physician will inject 2cc of the PL and 1cc of 0.5% ropivacaine into the epidural space. Once flow is confirmed for the epidural injection and facet with contrast, 1cc of the 14x PRP is injected into the facet joint. Procedure repeated on the opposite side and next level if indicated.
  Arms: PRP and PL Combo treatment

SUMMARY:
To evaluate and compare the effectiveness of 3 different injection treatments on multifidus atrophy and lower back pain.

DETAILED DESCRIPTION:
This study is a prospective, randomized controlled study of patients with atrophied multifidus muscles and axial lower back pain that are randomized to one of 3 treatment groups. Group 1 receives a series of 6 injections (1 time per week for 6 weeks) of platelet poor plasma into multifidus. Group 2 receives a series of 6 injections (1 time per week for 6 weeks) of platelet rich plasma (PRP) into multifidus. Group 3 receives a series of 3 injections (1 time every 2 weeks for 6 weeks) of PRP to multifidus, as well as PRP into facet joint, as well as an epidural injection of platelet lysate (PL).

Prior to procedure patient will undergo evaluation of medical history, back pain history, lumbar examination, medication use and review MRI of lumbar spine.

While lying prone, the patient's back will be exposed and prepped sterilely. While maintaining sterile technique, the physician will utilize US, x-ray or a combination of the two to guide the needles bilaterally into the multifidus, specifically the area of treatment using ultrasound, x-ray or a combination of the two. Once the lamina is reached the physician will either inject autologous 2.5 cc PPP (group 1) or will inject autologous 2.5 cc of 5x PRP into the multifidus muscle on one side and then repeat this on the opposite side for each level (group 2 & 3).

Additionally, for patients in group 3, using sterile technique under fluoroscopic guidance, the physician will guide a needle into the supraneural transforaminal space to perform an epidural injection with 2cc of 3x PL and 1 cc of 0.5% ropivacaine. Next, a needle will then be guided into the facet joint to perform an intra-articular injection with 1cc of 14x PRP. After the procedure, the patient will be cleaned and bandaged. The patient will be given standard rehab protocols to perform at home.

Patients will have follow-up visits with patient reported outcomes or pain and function at 3 months, 6 months and 12 months. A post-treatment MRI at 6 months will be compared to baseline MRI to measure changes to multifidus atrophy.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary signature of the Informed Consent
2. Axial low back pain for a minimum of 3 months
3. Male or female ages 18-75
4. Recent MRI (within last 6 months) consistent Kader grade 2 or 3 multifidus atrophy at 1 or 2 levels
5. Is independent, ambulatory, and can comply with all post-operative evaluations and visits

Exclusion Criteria:

1. Mild multifidus atrophy Kader grade 1
2. Multifidus atrophy at more than 2 levels
3. Symptomatic spinal stenosis (e.g. pseudoclaudication with moderate or severe MRI findings of stenosis)
4. Radicular symptoms (e.g. lower extremity radiating numbness, tingling, paresthesia, etc)
5. Fracture, previous spine surgery, neuromuscular disease of the trunk, malignancy, infection, or pregnancy
6. Radiofrequency ablation within the previous 12 months
7. Corticosteroid injection (epidural or facet) within the past 3 months
8. Contraindications for MRI
9. Condition represents a worker's compensation case
10. Currently involved in a health-related litigation procedure
11. Bleeding disorders
12. Allergy or intolerance to study medication
13. Use of chronic opioid
14. Documented history of drug abuse within six months of treatment
15. Any other condition, that in the opinion of the investigator, that would preclude the patient from enrollment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-06-29 (Actual)

PRIMARY OUTCOMES:
Post-treatment MRI | 6 months
  Change in multifidus atrophy from baseline MRI

SECONDARY OUTCOMES:
Single Assessment Numeric Evaluation Improvement Rating-modified | 3 months, 6 months, 12 months
  Difference between groups for mean improvement scores where -100=100% worse from baseline and 100=100% improved from baseline
Numeric Pain Scale | 3 months, 6 months, 12 months
  Difference between groups for numeric pain scores where 0=no pain and 10=worst pain possible
Functional Rating Index | 3 months, 6 months, 12 months
  Difference between groups for function scores where 0=minimal disability and 100=severe disability
Oswestry Low Back Disability Index | 3 months, 6 months, 12 months
  Difference between groups for function scores where 0=minimal disability and 100=severe crippling disability

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Centeno, MD, Principal Investigator — Centeno-Schultz Clinic
Locations (2):
- United States (2):
  - Centeno-Schultz Clinic, Broomfield, Colorado
  - Centeno-Schultz Clinic, Lone Tree, Colorado

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aure OF, Nilsen JH, Vasseljen O. Manual therapy and exercise therapy in patients with chronic low back pain: a randomized, controlled trial with 1-year follow-up. Spine (Phila Pa 1976). 2003 Mar 15;28(6):525-31; discussion 531-2. doi: 10.1097/01.BRS.0000049921.04200.A6. PMID 12642755
- [Background] Suni J, Rinne M, Natri A, Statistisian MP, Parkkari J, Alaranta H. Control of the lumbar neutral zone decreases low back pain and improves self-evaluated work ability: a 12-month randomized controlled study. Spine (Phila Pa 1976). 2006 Aug 15;31(18):E611-20. doi: 10.1097/01.brs.0000231701.76452.05. PMID 16915076
- [Background] Freeman MD, Woodham MA, Woodham AW. The role of the lumbar multifidus in chronic low back pain: a review. PM R. 2010 Feb;2(2):142-6; quiz 1 p following 167. doi: 10.1016/j.pmrj.2009.11.006. PMID 20193941
- [Background] Hodges PW, James G, Blomster L, Hall L, Schmid A, Shu C, Little C, Melrose J. Multifidus Muscle Changes After Back Injury Are Characterized by Structural Remodeling of Muscle, Adipose and Connective Tissue, but Not Muscle Atrophy: Molecular and Morphological Evidence. Spine (Phila Pa 1976). 2015 Jul 15;40(14):1057-71. doi: 10.1097/BRS.0000000000000972. PMID 25943090
- [Background] Kader DF, Wardlaw D, Smith FW. Correlation between the MRI changes in the lumbar multifidus muscles and leg pain. Clin Radiol. 2000 Feb;55(2):145-9. doi: 10.1053/crad.1999.0340. PMID 10657162
- [Background] Hussein M, Hussein T. Effect of autologous platelet leukocyte rich plasma injections on atrophied lumbar multifidus muscle in low back pain patients with monosegmental degenerative disc disease. SICOT J. 2016 Mar 22;2:12. doi: 10.1051/sicotj/2016002. PMID 27163101
- [Background] Sicari BM, Agrawal V, Siu BF, Medberry CJ, Dearth CL, Turner NJ, Badylak SF. A murine model of volumetric muscle loss and a regenerative medicine approach for tissue replacement. Tissue Eng Part A. 2012 Oct;18(19-20):1941-8. doi: 10.1089/ten.TEA.2012.0475. PMID 22906411
- [Background] Miroshnychenko O, Chang WT, Dragoo JL. The Use of Platelet-Rich and Platelet-Poor Plasma to Enhance Differentiation of Skeletal Myoblasts: Implications for the Use of Autologous Blood Products for Muscle Regeneration. Am J Sports Med. 2017 Mar;45(4):945-953. doi: 10.1177/0363546516677547. Epub 2016 Dec 27. PMID 28027451
- [Background] Gentile NE, Stearns KM, Brown EH, Rubin JP, Boninger ML, Dearth CL, Ambrosio F, Badylak SF. Targeted rehabilitation after extracellular matrix scaffold transplantation for the treatment of volumetric muscle loss. Am J Phys Med Rehabil. 2014 Nov;93(11 Suppl 3):S79-87. doi: 10.1097/PHM.0000000000000145. PMID 25133624